CLINICAL TRIAL: NCT03088826
Title: Comparison of Analgesic Efficacy of Morphine Sulfate Immediate Release (MSIR)/Acetaminophen vs. Oxycodone/Acetaminophen (Percocet) for Acute Pain in Emergency Department Patients
Brief Title: Analgesic Efficacy of (MSIR)/Acetaminophen vs. Oxycodone/Acetaminophen (Percocet)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Co-Investigator, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-01-05
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-08

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Morphine; Oxycodone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSIR and Acetaminophen Group (Active Comparator): The patients in this group will receive 1 tablet 15mg PO morphine sulfate immediate release combined with 650mg of Acetaminophen
  Interventions: Drug: Morphine Sulfate; Drug: Acetaminophen
- Oxycodone and Acetaminophen Group (Active Comparator): The patients in this group will receive 1 tablet 10mg Oxycodone combined with 650mg of Acetaminophen
  Interventions: Drug: Oxycodone; Drug: Acetaminophen

INTERVENTIONS:
Drug: Morphine Sulfate — 15mg PO morphine sulfate
  Arms: MSIR and Acetaminophen Group
Drug: Oxycodone — 10mg Oxycodone
  Arms: Oxycodone and Acetaminophen Group
Drug: Acetaminophen — 650 mg Acetaminophen

SUMMARY:
Oxycodone and Hydrocodone are the most commonly used oral opioid analgesics in the emergency department and in outpatient settings. Both medications have a very high potential for abuse due to the prominence of the euphoric effect (abuse liability) and relative lack of "bad "or "negative" effects (likeability). The highly addictive properties of these medications lead to recurrent ED visits for repetitive dosing and prescribing that may lead to abuse, misuse, development of dependence and addiction, and, most importantly, death due to overdose. In contrast, several research papers demonstrated that administration of MSIR results in similar analgesic efficacy to Oxycodone and Hydrocodone but with significantly less euphoric and rewarding associated effects. In addition, consumption of large doses of MSIR leads to dysphoria, vomiting and sedation ("negative effects"). To the investigators' knowledge, there are no randomized controlled trials in the ED that directly compared analgesic efficacy of MSIR to Percocet

DETAILED DESCRIPTION:
The investigators' hypothesis is that MSIR coupled with acetaminophen will have similar if not better analgesic efficacy at 30 minutes and 1 hour than oxycodone coupled with acetaminophen for acute painful conditions in the emergency department.

This study will be a double-blind randomized clinical trial evaluation analgesic efficacy of orally administered MISIR+acetaminophen in comparison to Oxycodone+acetaminophen for treating pain. Patients will be enrolled from a single ED in a tertiary academic center.

Patients based on inclusion criteria will be randomized to receive either 1 tablet of 15mg PO morphine sulfate immediate release combined with 650mg of Acetaminophen or 1 tablet 10mg Oxycodone combined with 650 mg Acetaminophen. All drugs will be crushed and given to the subjects in blinded fashion. Patients, physicians, nurses and research assistants will be blinded to drug assignment throughout the study. Medication will be prepared by on site pharmacist.

Pain will be reassessed at both 30 minutes, 45 minutes and 1 hour with the primary outcome of reduction in pain score by 1.3 points at 60 minutes. Assuming a 1.7 pain difference is minimally significant clinically with standard deviation of 3.0 (based on a previous study of morphine analgesia), a minimum of 50 patients per group will be needed for 80% power with alpha equal to 0.05.

Secondary outcomes will include any reported adverse effects; the requirement of additional analgesia.

Generalized likability and chance of repeated use will be reported by using a visual analogue scale with following questions:

"Do you feel any DRUG EFFECT?" "Do you LIKE the drug?" "How HIGH are you?" "Does the drug have any GOOD EFFECTS?" "Does the drug have any BAD EFFECTS?" "How much do you DESIRE the medication?" " Does the drug make you have UNPLEASANT THOUGHTS?" "Does the drug make you have UNPLEASANT BODILY SENSATIONS?" "Does the drug make you feel IRRITATED?" "Does the drug make it DIFFICULT TO CONCENTRATE?"

The patients will respond by positioning an arrow along a 100-point line labeled with "not at all" at one end and "extremely" at the other.

Data will be analyzed by intention to treat and will include frequency distributions, and Student's T-test to assess a difference in pain scores and vital signs. The chi-square test will assess the presence or absence of side effects between the two groups. Statistical analyses will be conducted by the research manager and the hospital senior biostatistician who will be independent of all data collection.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-64,
* present to the Emergency department with moderate-to-severe acute pain that warrants an oral opioid analgesic.
* pain score is above 5 and are deemed to require oral opioid at the discretion of the attending physician.
* Painful conditions will include but will not be limited to acute traumatic/non-traumatic musculoskeletal pain, renal colic pain, dental pain.

Exclusion Criteria:

* age <18, age >64,
* subjects who received long acting opioids within 24 hours of presenting to ED
* received short acting analgesics within 4 hours,
* chronic pain,
* pregnant patients,
* patient refusal,
* altered mental status,
* known allergy to either morphine or oxycodone or acetaminophen,
* history of substance and opioid abuse,
* unstable vital signs, acute psychosis or incarceration.
* subjects who received long acting opioids within 24 hours of presenting to ED;
* chronic pain"

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MSIR and Acetaminophen Group | Oxycodone and Acetaminophen Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSIR and Acetaminophen Group | Oxycodone and Acetaminophen Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (13.2) | 46.3 (14.6) | 43.5 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 20 | 32
  Male | 28 | 20 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Pain Reduction at 60 Minutes (Baseline Pain Score - Pain Score at 60 Minutes)
Description: The reduction of pain at 60 minutes from baseline: The pain scale ranges from 0 to 10 with 0 being no pain, 5 being moderate pain and 10 being very severe pain.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSIR and Acetaminophen Group | Oxycodone and Acetaminophen Group
Number analyzed (Participants) | 40 | 40
units on a scale | 3.95 (2.29) | 3.95 (2.37)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | MSIR and Acetaminophen Group | Oxycodone and Acetaminophen Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03088826/Prot_SAP_000.pdf